CLINICAL TRIAL: NCT02589236
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of N91115 to Evaluate Efficacy and Safety in Patients With Cystic Fibrosis Who Are Homozygous for the F508del-CFTR Mutation Treated With Lumacaftor/Ivacaftor
Brief Title: Study of Cavosonstat (N91115) in Patients With CF Homozygous for the F508del-CFTR Mutation
Acronym: SNO-6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Collaborators: Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N91115-2CF-05
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; N91115; Cavosonstat
MeSH Terms: conditions — Cystic Fibrosis | interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo Capsule
  Interventions: Drug: Placebo
- Cavosonstat (N91115) 200 mg (Experimental): Cavosonstat (N91115) 200 mg twice daily (BID)
  Interventions: Drug: Cavosonstat
- Cavosonstat (N91115) 400 mg (Experimental): Cavosonstat (N91115) 400 mg BID
  Interventions: Drug: Cavosonstat

INTERVENTIONS:
Drug: Cavosonstat — GSNOR inhibitor
  Other Names: N91115
  Arms: Cavosonstat (N91115) 200 mg; Cavosonstat (N91115) 400 mg
Drug: Placebo — Control sample with only capsule excipients and fillers
  Other Names: control
  Arms: Placebo

SUMMARY:
This will be a double-blind, randomized, placebo-controlled, parallel group study. The purpose of this study is to investigate the efficacy and safety of Cavosonstat (N91115) in adult patients with CF who are homozygous for the F508del-CFTR mutation and being treated with lumacaftor/ivacaftor (Orkambi™).

DETAILED DESCRIPTION:
Primary Objective:

* Assess the efficacy of N91115 at 12 weeks when added to preexisting treatment with lumacaftor/ivacaftor in adult patients with CF who are homozygous for the F508del-CFTR mutation

Secondary Objectives:

* Assess the effect of N91115 added to lumacaftor/ivacaftor on safety
* Assess the effect of lumacaftor/ivacaftor added to N91115 on the pharmacokinetics of N91115, lumacaftor, and ivacaftor

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been treated with lumacaftor/ivacaftor for at least 8 weeks prior to Day 1 (start of dosing)
* A history of Sweat Chloride (SC) ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT) (either before or after starting lumacaftor/ivacaftor treatment)
* Body weight ≥ 40 kg
* ppFEV1 40 - 85 % predicted (inclusive) at screening
* Oxygen saturation ≥ 90% breathing ambient air at screening

Exclusion Criteria:

* Any acute infection that requires treatment or hospitalization within 2 weeks of Study Day 1
* Colonization with organisms associated with more rapid decline in pulmonary status, such as Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus
* Any change in the regimen for chronic therapies for CF lung disease (e.g., Pulmozyme®, hypertonic saline, Azithromycin, TOBI®, Cayston®) within 4 weeks of Study Day 1
* Are pregnant, planning a pregnancy, or breast-feeding at screening
* Blood hemoglobin < 10 g/dL at screening
* Serum albumin < 2.5 g/dL at screening
* Abnormal liver function defined as ≥ 3 x upper limit of normal (ULN)
* History of abnormal renal function within 3 months of screening
* History of ventricular tachycardia or other clinically significant ventricular arrhythmias
* History, including the screening assessment, of prolonged QT and/or QTcF (Fridericia's correction) interval
* History of solid organ or hematological transplantation
* History of alcohol abuse or drug abuse
* Ongoing participation in another therapeutic clinical trial
* Use of continuous (24 hr/day) or nocturnal supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in percent predicted FEV1 (ppFEV1) | From baseline to 12 weeks
  Forced Expiratory Volume in one second (FEV1) from before study (Baseline) to after 12 weeks of N91115 treatment

SECONDARY OUTCOMES:
Relative change from baseline in ppFEV1 | baseline to 12 weeks
  Forced Expiratory Volume in one second (FEV1) from before study (Baseline) to after 12 weeks of N91115 treatment
Absolute change from baseline in sweat chloride | baseline to 12 weeks
  A sweat chloride measurement on the skin at study start and after 12 weeks of N91115
Absolute change from baseline in Cystic Fibrosis Questionnaire -Revised CFQ-R (respiratory symptom scale) | baseline to 16 weeks
  Comparison of the Questionnaire from study start to 16 weeks
Absolute change from baseline in body mass index (BMI) | baseline to 12 weeks
  Assessment of change in body mass index from study start to after 12 weeks of N91115
Absolute change from baseline in Patient Global Impression of Change (PGIC) | baseline to 12 weeks
  Patient reported outcome journal
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | baseline to 16 weeks
  Any adverse events assessment including clinical laboratory values, electrocardiogram (ECG), pulmonary exacerbations, or vital sign changes
Pharmacokinetic Measurements of Maximum Plasma Concentration [Cmax], of N91115, lumacaftor, and ivacaftor | baseline to 12 weeks
  Maximum Plasma Concentration [Cmax] measurements of N91115, lumacaftor and ivacaftor
Pharmacokinetic Measurements of Area Under the Curve (AUC) for N91115, Ivacaftor and lumacaftor | baseline to 12 weeks
  AUC measurements of N91115, lumacaftor and ivacaftor

OTHER OUTCOMES:
Number of pulmonary exacerbations | baseline to 12 weeks
  Assessment of number of pulmonary exacerbations at baseline compared through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (46):
- United States (46):
  - University of Alabama, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Via Christi Research, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Wayne State University-Harper, Detroit, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital - Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - ProMedica Toledo Children's Hospital, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Hospital | Austin Children's Chest Associates, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical Center of Wisconsin, Madison, Wisconsin